CLINICAL TRIAL: NCT06317792
Title: Assessing the Efficacy of Online Exergaming-Integrated Physiotherapy for Parkinson's Disease: A Validation Study
Brief Title: The Efficacy of Online Exergaming-Integrated Physiotherapy for Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cheng-Hsien Lu, MD, MSc, Professor of neurology, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202201719B0
Record Dates: First submitted 2024-02-21; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Parkinsonism in Diseases Classified Elsewhere
Keywords: online exergaming-based physiotherapy; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups in a randomized controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online exergaming-based physiotherapy intervention group (Experimental): The training tasks consist of a set of 10 pieces of training (20 min per session, five sessions every week, for 8 weeks)
  Interventions: Other: online exergaming-based physiotherapy programs
- Online exergaming-based physiotherapy observation group (No Intervention): Observation only

INTERVENTIONS:
Other: online exergaming-based physiotherapy programs — The online exergaming-based physiotherapy programs focus on training in shoulder, hip, and knee ROM balance, weight-bearing, strength, weight shifting, and walking based on RF in machine learning to the features selection in patients with PIGD. The training tasks consist of a set of 10 pieces of training (20 min per session, five sessions every week, for 8 weeks). Five exergaming programs were used for training, designed to incorporate an appropriate level of challenge to match the ability and fitness of patients with PD.
  Arms: Online exergaming-based physiotherapy intervention group

SUMMARY:
To validate the efficiency of online exergaming-based physiotherapy. We will enroll patients with Parkinson's disease in postural instability and gait disturbance motor phenotype in the study and divide them into two groups in a randomized controlled study.

DETAILED DESCRIPTION:
The investigators will enroll patients in PIGD and divide them into two groups in a randomized controlled study. Participants received an exergaming intervention using the Kinect sensor (Microsoft Corporation, Redmond, WA, USA) from a commercially available exercise system (HappyGoGo, LONGGOOD MEDITECH LTD., Taipei, Taiwan). The Kinect sensor incorporates infrared light and a video camera, which creates a 3D map of the area in front of it. This device provides full-body 3D motion capture.

The online exergaming-based physiotherapy programs focus on training in shoulder, hip, and knee ROM balance, weight-bearing, strength, weight shifting, and walking based on RF in machine learning to the features selection in patients with PIGD. The training tasks consist of 10 pieces of training (20 minutes per session, five sessions every week, for 8 weeks). Five exergaming programs were used for training, designed to incorporate an appropriate level of challenge to match the ability and fitness of patients with PD.

To confirm the status of individual training at home, the data will be sent back to the computer output report of the medical side after each training is completed. These data include the quantitative data of a joint ROM, the movement cycle change diagram, and the upper and low limb movements decomposed by each movement plane. The investigators also obtain the trajectory path mapping to understand whether the quality of individual actions is accurate, in place, and line with expected benchmarks.

Safety and Tolerability: If the patient can not complete half of the rehabilitation program, this/her data will be excluded from the analysis.

Exergame rehabilitation outcome assessments To evaluate the efficiency and the durability of the training effect. Outcomes were measured at five different periods including Month 0 (pretest) (clinical score, gait cycle, cognitive function, and fMRI), Month 2 (posttest) (clinical score, gait cycle, and fMRI), and Month 8 (follow-up) (clinical score, gait cycle, and cognitive function) and Year 2 and year 3 (follow-up) (clinical score, gait cycle, and cognitive function).

1. Functional Outcome Measure: Clinical scores and parameters of walking gait cycle The Functional Outcome measure includes the (1) UPDRS score, (2) Tinetti balance and gait score, (3) Berg Balance Scale, (4) Time-up to go test, and (5) parameters in the gait cycle including plantar pressure measurement, static and dynamic balance measures, COP trajectory measurements during gait initiation, and spatiotemporal and kinematic gait analysis in straightforward walking and turning through study completion, an average of three years.
2. Secondary outcome measures include Severity, frequency, and situations of falling and Physical (balance, mobility, freezing of gait, habitual physical activity) and psychological (fear of falling, affect) measures during the intervention and through study completion, an average of three years.

ELIGIBILITY:
Inclusion Criteria:

1． Clinical diagnosis of Parkinson's disease

Exclusion Criteria:

1. Moderate and severe dementia (Clinical Dementia Rating more than or equal to 2)
2. Advanced PD stage (Hoehn and Yahr staging equal or more than four)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale score assessment | Intervention and follow-up period through study completion, an average of 3 years
  The outcome measure is the Unified Parkinson's Disease Rating Scale score. The UPDRS scale consists of the following six segments: 1) Mentation, Behavior, and Mood, 2) ADL, 3) Motor sections, and 4) Complications of Therapy (in the past week) The four segments are made up of 42 items grouped into four subscales. Each item has 0-4 ratings: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe)
Tinetti balance and gait score assessment | Intervention and follow-up period through study completion, an average of 3 years
  The score consists of two parts, including the balance score (score=0-16) and gait score (score=0-12), and ranged from 0 to 28 points by summing the points obtained for each of the two tests.

SECONDARY OUTCOMES:
Fall Risk assessment using Berg Balance Scale | intervention and follow-up period through study completion, an average of 3 years
  The maximum obtainable Berg Balance Scale is 56 and there are four ranges of scores. Patients scoring range of 41-56, 21-40, and 0 -20 indicate low fall risk, medium fall risk, and high fall risk, respectively
Depression severity assessment | intervention and follow-up period through study completion, an average of 3 years
  To obtain a patient-based measurement of depression, the Geriatric Depression Scale (GDS-30) was used. Depression severity was classified using the GDS-30 as follows: No depression (GDS 0-9), mild depression (GDS 10-19), and severe depression (GDS 20-30).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Chang Gung University College of Medicine, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR